CLINICAL TRIAL: NCT01144390
Title: Barriers and Effect of Optimizing Intervention Protocols for Heroin Dependence in Community-based Methadone Maintenance Treatment (MMT): a Cohort Study
Brief Title: Effect Study of Optimized Intervention to Heroin Addicts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Min ZHAO, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiMHC
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Heroin Dependence
Keywords: heroin dependence; community-based; MMT
MeSH Terms: conditions — Heroin Dependence | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CBT plus MMT (Experimental): cognitive behavioral therapy for heroin addicts with methadone maintenance treatment
  Interventions: Behavioral: cognitive behavioral therapy; Drug: methadone maintenance treatment
- methadone maintenance treatment (Active Comparator): methadone maintenance treatment for heroin addicts
  Interventions: Drug: methadone maintenance treatment

INTERVENTIONS:
Behavioral: cognitive behavioral therapy — cognitive behavioral therapy, one session per week and psycho-education lecture in group once per month
  Arms: CBT plus MMT
Drug: methadone maintenance treatment — methadone maintenance treatment

SUMMARY:
The purpose of this study is to explore barriers and determine whether optimizing protocol is effective in the treatment of heroin dependence in community-based MMT clinics.

DETAILED DESCRIPTION:
Drug dependence is one of the most serious public health problems worldwide. In China, among more than 100, 0000 registered drug addicts mostly are heroin dependence. Drug dependence post great risks to physical condition, their family and society, and can lead to infectious disease transmission. Though almost 500 MMT clinics which can offer MMT service to heroin addicts have been set up, there are still some problems, for example, poor compliance, high rate of dropping out and relapse which affect the service delivery to them. The guideline developed by WHO focused on psychotherapy to opiate addicts with MMT. So delivery of a set of comprehensive, integrated psychotherapy to opiate addicts is very critical in such methadone clinics.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of heroin dependence
* must be able to take methadone

Exclusion Criteria:

* schizophrenia and mood disorder
* physical disabilities who could not come to take part in psychotherapy sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2010-04; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
treatment retention | 12 months
  retaining patients in the methadone maintenance treatment during and after the study.

SECONDARY OUTCOMES:
in-treatment performance. | 12 months
  treatment performance of addicts include: treatment sessions during the study, negative urine specimens, drop-out rate, severity of ASI,scores of HIV-related high risk sexual behavior, the temperature and character inventory, perceived stigma scale, self-esteem inventory,self efficacy, social support scores,drug use from self-report from baseline to 3 month and 6 month.

CONTACTS AND LOCATIONS:
Overall Officials: min ZHAO, Ph.D., Principal Investigator — Shanghai Mental Health Center
Locations (4):
- China (4):
  - Mental Health Center of Hongkou District, Shanghai, Shanghai Municipality
  - Mental Health Center of Pudong District, Shanghai, Shanghai Municipality
  - Mental Health Center of Xuhui District, Shanghai, Shanghai Municipality
  - Mental Health Center of Yangpu District, Shanghai, Shanghai Municipality

REFERENCES:
- [Derived] Pan S, Jiang H, Du J, Chen H, Li Z, Ling W, Zhao M. Efficacy of Cognitive Behavioral Therapy on Opiate Use and Retention in Methadone Maintenance Treatment in China: A Randomised Trial. PLoS One. 2015 Jun 24;10(6):e0127598. doi: 10.1371/journal.pone.0127598. eCollection 2015. PMID 26107818